CLINICAL TRIAL: NCT03450577
Title: International Prospective Register on Treatment of Coronary Artery Bifurcation Lesions
Brief Title: International Bifurcation Study
Acronym: IBS
Status: Recruiting | Type: Observational
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Dmitrii Khelimskii, Dmitrii Khelimskii, Meshalkin Research Institute of Pathology of Circulation
Other Study IDs: IBS
Record Dates: First submitted 2018-02-05; First posted 2018-03-01 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Coronary Bifurcation Lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCI of bifurcation lesions: Patients who have undergone bifurcation coronary artery stenting.
  Interventions: Procedure: PCI of bifurcation lesions

INTERVENTIONS:
Procedure: PCI of bifurcation lesions — Different approaches for treatment of bifurcation coronary artery disease.

SUMMARY:
The IBS registry is an observational, multi-center, real-world registry of stenting in coronary bifurcation lesions that will collect information on procedures and outcomes from various participating centers.

The aim of this registry is to investigate long-term clinical results and predictors of adverse outcomes after PCI for coronary bifurcation lesions among various participating centers.

DETAILED DESCRIPTION:
Patients with coronary bifurcation lesions, if they meets all the study inclusion criteria and none of the exclusion criteria, after signing the informed consent, they will underwent PCI according to the current standard of care and will be entered in the registry. Follow-up for all subjects will continue for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Any type of bifurcation lesion in major epicardial artery

Exclusion Criteria:

* Patient refused informed consent to participate in the registry

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary bifurcation lesion treated during PCI
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedural success | 1 day
  Achievement of technical success and with no in-hospital major adverse cardiac events

SECONDARY OUTCOMES:
Major Adverse Cardiac and Cerebrovascular Events | 6 months, 1 year, 3 years, 5 years
  Death, myocardial infarction (MI), target vessel revascularization (TVR), or stroke.
All cause mortality | 6 months, 1 year, 3 years, 5 years
  All of the deaths that occur in a study group, regardless of the cause.
Death from cardiac causes | 6 months, 1 year, 3 years, 5 years
  All deaths will be assumed cardiovascular in nature unless a non-cardiovascular cause can be clearly provided (e.g. malignancy, trauma, and infection).
Myocardial infarction | 6 months, 1 year, 3 years, 5 years
  The presence of electrocardiography findings indicative of ischemia that were not related to the index procedure, as well as chest discomfort associated with creatinine kinase-myocardial band fraction or troponin-T/troponin I greater than the upper limit of normal.
Target vessel revascularization | 6 months, 1 year, 3 years, 5 years
  Repeat PCI of the lesion within 5 mm of stent deployment or bypass graft surgery of the target vessel.
Stent thrombosis | 6 months, 1 year, 3 years, 5 years
  Sudden occlusion of a stented coronary artery due to formation of thrombosis.According to the Academic Research Consortium was defined as definite, probable, or possible.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitrii Khelimskii, MD, Principal Investigator — Meshalkin National Medical Research Center
Locations (1):
- Meshalkin National Research Center, Novosibirsk, Novosibirsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khelimskii D, Bessonov I, Sapozhnikov S, Badoyan A, Baranov A, Mamurjon M, Manukian S, Utegenov R, Krestyaninov O. Impact of Prolonged Dual Antiplatelet Therapy After Bifurcation Percutaneous Coronary Intervention in Patients with High Ischemic Risk. Am J Cardiovasc Drugs. 2024 Jul;24(4):577-588. doi: 10.1007/s40256-024-00657-1. Epub 2024 Jun 13. PMID 38871947
- See also: Related Info — http://meshalkin.ru